CLINICAL TRIAL: NCT01757145
Title: Eltrombopag for Enhancing Platelet Engraftment in Adult Patients Undergoing Cord Blood Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7114
Record Dates: First submitted 2012-12-06; First posted 2012-12-28 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2013-02

CONDITIONS: Hematological Malignancy; Bone Marrow Failure Syndrome
Keywords: Cord blood transplantation; Eltrombopag; Platelet engraftment
MeSH Terms: conditions — Hematologic Neoplasms; Bone Marrow Failure Disorders | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag will be given orally as a single daily dose. From day +1 after cord blood transplantation, start eltrombopag 100 mg/d. If primary end point not reached on day +14,then from day +15 - 150 mg/d. If primary end point not reached on day +28 then from day +29 - 200 mg/d. If primary end point not reached on day +42 then from day +43 and on - 300 mg/d (maximal dose). If dose not tolerated, return to last tolerated dose.
  Eltrombopag will be discontinued after platelet count has exceeded 50,000/microliter for 14 consecutive days without administration of platelets.
  In case of decline of platelet count < 30,000/microliter within 15 days from eltrombopag discontinuation, it will be resumed for additional 4 weeks.
  After 4 weeks we will re-attempt to hold the drug.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — From day +1, start eltrombopag 100 mg/d. If primary end point not reached on day +14, then from day +15 - 150 mg/d.
  If primary end point not reached on day +28 then from day +29 - 200 mg/d. If primary end point not reached on day +42 then from day +43 and on - 300 mg/d maximal dose).
  If present dose not tolerated, return to last tolerated dose. Eltrombopag will be discontinued after platelet count has exceeded 50,000/microliter for 14 consecutive days without administration of platelets. In case of decline of platelet count < 30,000/microliter within 15 days from eltrombopag discontinuation, it will be resumed for additional 4 weeks. After 4 weeks we will re-attempt to hold the drug (if the threshold of platelet count >50,000/microliter will be reached again).
  Other Names: Revolade

SUMMARY:
The purpose of this study is to determine whether Eltrombopag may shorten time to platelet engraftment after allogeneic cord blood transplantation.

DETAILED DESCRIPTION:
Platelet recovery is significantly hampered following umbilical cord blood (UCB) transplantation. Median time to platelet engraftment (defined as the first of 7 consecutive days of an unsupported platelet count of at least 20,000/microliter) in a large retrospective study was more than 70 days and cumulative incidence of platelet recovery at 6 months was 50.5%. In the pediatric population with acute leukemia median time to platelet engraftment with UCB transplantation was 59 days and cumulative incidence of platelet recovery at 6 months was 43%-73%, depending on human leukocyte antigen (HLA) disparity and cell dose. Recently, in a cohort of adult patients given myeloablative conditioning followed by double UCB transplantation, the cumulative incidence of platelet recovery (≥ 50,000/microliter)at 100 days was 53%. In another cohort of patients given reduced intensity conditioning regimen followed by single or double UCB transplantation, the median time to platelet recovery (≥ 50,000/microliter) and cumulative incidence of platelet recovery at 6 months were 49 days and 65%, respectively. Thus, after UCB transplantations, patients are platelet transfusion-dependent for prolong periods of time, resulting in many drawbacks, such as exposure to blood transfusions hazards, higher incidence of platelet allo-reactivity and extended periods of bleeding diathesis and undesirable costly and long hospitalizations.

Eltrombopag is a thrombopoietin-receptor agonist that initiates thrombopoietin-receptor signaling and thereby inducing proliferation and maturation of megakaryocytes.Administration of eltrombopag increased platelet production in volunteers with normal platelet counts, patients with thrombocytopenia secondary to hepatitis C virus infection and in patients with chronic immune thrombocytopenic purpura.

We will evaluate the safety and efficacy of eltrombopag treatment given early after UCB transplantation. The study is an open non-comparative study. The primary outcome will be cumulative incidence of partial platelet engraftment (first of 7 consecutive days of an unsupported platelet count of at least 20,000/microliter)at day 50 post transplantation. Secondary objectives are safety, tolerability and other transplantation related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 year old.
2. Patients receiving unmanipulated single or double umbilical cord blood allogeneic grafts.
3. Malignant and non malignant indications for transplantation.
4. Myeloablative and reduced intensity conditioning regimens.
5. Patients must meet all other pre-transplantation criteria of the transplantation center including acceptable tests of heart, liver, kidney, and lung function (standard screening for transplantation per PI, and co-investigators).
6. Able to give written informed consent for a clinical trial.
7. Able to comply with study protocol.

Exclusion Criteria:

1. Indications for transplantation

   1. Patients with primary myelofibrosis.
   2. M7 (French-American-British classification) acute myeloid leukemia. Acute leukemia secondary to a myeloproliferative neoplasm.
   3. Patients with persistent acute leukemia (>5% bone marrow blasts) at the time of transplantation.
2. Patients with prior thromboembolic event. Patients with previous catheter related thrombosis will be eligible if more than 3 months elapsed.
3. Hypersensitivity to eltrombopag.
4. Liver enzymes abnormalities:

   Alanine transaminase (ALT) levels > 3 times the upper limit of normal (ULN) or serum bilirubin > 1.5 ULN (unless due to Gilbert's syndrome or hemolytic bilirubin).
5. Pregnancy: Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation. A woman of child-bearing potential is defined as a woman who has not been naturally post-menopausal for at least 12 consecutive months or with no previous surgical sterilization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Platelet engraftment rate up to 50 days post transplantation, defined as the first of 7 consecutive days of an unsupported platelet count of at least 20,000/microliter. | 50 days

SECONDARY OUTCOMES:
Time to partial platelet engraftment, defined as the first of 7 consecutive days of an unsupported platelet count of at least 20,000/microliter. | 180 days
Time to sustained complete platelet engraftment defined as the first of 7 consecutive days of an unsupported platelet count of at least 50,000/microliter. | 180 days
Complete platelet engraftment rates up to 50 days post transplantation defined as the first of 7 consecutive days of an unsupported platelet count of at least 50,000/microliter. | 50 days
Time to neutrophil engraftment defined as the first of 3 consecutive days to achieve an absolute neutrophil count ≥ 500/microliter. | 60 days

OTHER OUTCOMES:
Any grade 3/4 adverse event | 12 months
  Number of participants with any grade 3/4 adverse event as a measure of safety and tolerability.
Thromboembolic events | 12 months
  Number of participants with a thromboembolic event as a measure of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Hadassah hospital, Jerusalem
  - Davidof Cancer Center, Beilinson hospital, Rabin medical center, Petah Tikva